CLINICAL TRIAL: NCT00132717
Title: An Open-Label, Multicenter Study to Assess the Efficacy of Switching to a Combination Tablet Ezetimibe/Simvastatin 10mg/40mg, Compared to Doubling the Dose of Statin in Patients Hospitalized With a Coronary Event
Brief Title: A 12 Week Study of MK0653A in Patients Who Have Been Hospitalized for a Possible Heart Problem (0653A-808)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-808; 2004_046
Record Dates: First submitted 2005-08-02; First posted 2005-08-22 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Simvastatin

INTERVENTIONS:
Drug: MK0653A (ezetimibe [+] simvastatin)
Drug: Comparator: atorvastatin
Drug: Comparator: fluvastatin
Drug: Comparator: lovastatin
Drug: Comparator: pravastatin
Drug: Comparator: rosuvastatin
Drug: Comparator: simvastatin

SUMMARY:
The purpose of this study is to investigate the effect of an investigational cholesterol-lowering drug in patients who are currently taking an approved medication for hypercholesterolemia (high cholesterol levels) and have been hospitalized for a heart problem.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years old, who were admitted to a hospital for an investigation of a heart problem and are currently receiving an approved medication to lower cholesterol

Exclusion Criteria:

* Patients who have congestive heart failure (CHF), uncontrolled high blood pressure, poorly controlled blood sugar, impaired kidney function, or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2007-06-01 (Actual); Study Completion 2007-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of MK0653A compared to doubling the statin dose as shown by the low-density lipoprotein cholesterol (LDL-C) values achieved after 12 weeks of treatment | After 12 weeks of treatment

SECONDARY OUTCOMES:
To determine the effect of MK0653A compared to doubling the statin dose on total cholesterol (TC) after 12 weeks | After 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Reckless JP, Henry P, Pomykaj T, Lim ST, Massaad R, Vandormael K, Johnson-Levonas AO, Lis K, Brudi P, Allen C. Lipid-altering efficacy of ezetimibe/simvastatin 10/40 mg compared with doubling the statin dose in patients admitted to the hospital for a recent coronary event: the INFORCE study. Int J Clin Pract. 2008 Apr;62(4):539-54. doi: 10.1111/j.1742-1241.2008.01697.x. Epub 2008 Feb 11. PMID 18266852
- [Background] Brudi P, Reckless JP, Henry DP, Pomykaj T, Lim ST, Massaad R, Vandormael K, Johnson-Levonas AO. Efficacy of ezetimibe/simvastatin 10/40 mg compared to doubling the dose of low-, medium- and high-potency statin monotherapy in patients with a recent coronary event. Cardiology. 2009;113(2):89-97. doi: 10.1159/000172795. Epub 2008 Nov 15. PMID 19018143